CLINICAL TRIAL: NCT06150885
Title: A Single Arm, Open Label, Dose-escalation Phase I and Dose-expansion Phase IIa Clinical Study to Evaluate the Feasibility, Safety, and Efficacy of Allogeneic Chimeric Antigen Receptor (CAR) Gamma-Delta T Cells CAR001 in Subjects with Relapsed/refractory Solid Tumors
Brief Title: A Safety and Efficacy Study of Allogeneic CAR Gamma-Delta T Cells in Subjects with Relapsed/Refractory Solid Tumors
Acronym: CAR001
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ever Supreme Bio Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-CCAR01-A3301
Record Dates: First submitted 2023-11-13; First posted 2023-11-29 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR001 (Experimental): CAR001 cells mixed with normal saline will be administered to patients.
  Interventions: Biological: HLA-G-CAR.BiTE allogeneic γδ T cells

INTERVENTIONS:
Biological: HLA-G-CAR.BiTE allogeneic γδ T cells — Phase I is a multiple escalating dose, single arm, open-label and 3+3 design that implemented with five cohorts: low dose for single administration, low dose for twice administrations for 2 weeks, low, middle and high dose for 4 repeated administrations for 4 weeks.
  Phase IIa is a single-arm, open-label and dose-expansion study and the effective dose of CAR-positive cells will be administered to 27 evaluable subjects with TNBC, NSCLC, CRC or GBM via intravenous infusion weekly for 4 weeks.

SUMMARY:
This study is composed of phase I and IIa parts. The dose-escalation phase I part aims to find the maximum tolerated dose (MTD) and to identify the safety of CAR001 in subjects with relapsed/refractory solid tumor; the dose-expansion phase IIa part aims to evaluate the potential efficacy of CAR001 in subjects with relapsed/refractory non-small cell lung cancer (NSCLC), triple negative breast cancer (TNBC), colorectal cancer (CRC) or Glioblastoma multiforme (GBM).

DETAILED DESCRIPTION:
Primary Objective:

Phase I:

To evaluate the safety of CAR001 in subjects.

Phase IIa:

To provide potential evidence for the clinical efficacy of CAR001 in improving tumor response rate in subjects.

Secondary Objectives:

To evaluate the safety and potential efficacy of CAR001 in subjects.

Exploratory:

Level of CAR-positive γδT cells in peripheral blood from baseline to subsequent visits. (Time Frame: 12 months after the last infusion)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years
2. For phase I part, subjects with histologically confirmed diagnosis of solid tumor with expression of PD-L1 ≥ 1% and are relapsed/refractory to at least two lines of standard-of-care therapy. For phase IIa part, subjects with histologically confirmed diagnosis of TNBC, NSCLC, CRC or GBM with expression of PD-L1 ≥ 1%, and are relapsed/refractory to at least two lines of standard-of-care therapy.
3. With at least one measurable lesion as defined by RECIST1.1 (for TNBC, NSCLC or CRC) or RANO (for GBM)
4. Able to understand and sign the ICF
5. Have a life expectancy of > 12 weeks
6. ECOG performance status ≤ 1
7. Recovered from any previous therapy related toxicity to ≤ grade 2 at screening
8. With adequate renal function: serum creatinine ≤ 1.5 X ULN; eGFR > 50 ml/min
9. With adequate liver function: ALT, AST, and ALP ≤ 3X ULN or ≤ 5 X ULN if liver metastases; and total bilirubin ≤ 1.5X ULN or ≤ 3 X ULN if due to Gilbert's disease
10. With PT and PTT ≤ 1.5X ULN
11. With adequate hematopoietic function:

    * ANC ≥ 1,000 cells/μl
    * Platelets ≥ 75,000 counts/μl
    * Total WBC ≥ 2,000 cells/μl
    * Hemoglobin ≥ 8 g/dL

Exclusion Criteria:

1. Has received any allogeneic cell therapy before screening
2. With known or suspected to be hypersensitivity to CAR001 or its excipients, such as DMSO or human serum albumin
3. With more than one kind of active diagnosed primary cancer
4. With active infection requiring systemic medication
5. With medical conditions who are receiving systemic steroid therapy >10 mg prednisone/day or equivalent dose, or other immune-suppressants in the past 2 weeks
6. Has been diagnosed as HIV positive (confirmed by anti-HIV and nucleic acid test)
7. With acute cardiovascular disease; NYHA classification ≥ 3; or history of myocardial infarction during the past 6 months; or has active uncontrolled arterial hypertension by medical history. Per investigator's judgment, would not make participation appropriate
8. With historical or current auto-immune diseases, such as rheumatoid arthritis, type I diabetes, psoriasis or systemic lupus erythematosus
9. Has uncontrolled psychiatric disorder by medical history
10. Has CNS diseases except GBM or stroke
11. Has received any investigational therapy from another clinical study within 4 weeks
12. Inability to undergo radiological assessment, such as MRI or CT for any reason
13. Has received radiotherapy or chemotherapy within 2 weeks (but palliative radiation therapy (R/T) for pain control are allowed)
14. Not suitable to participate the trial as judged by the investigator
15. Female subject of childbearing potential who:

    * Is lactating; or
    * Has a positive pregnancy test result at eligibility checking; or
    * Refuses to adopt at least two form of birth control from signing informed consent to 1 year after the last administration of CAR001.
16. Male subject with a female spouse/partner who is of childbearing potential refuses to adopt at least two forms of birth control from signing informed consent to 1 year after the last administration of CAR001.

For exclusion criteria #15 and #16, acceptable forms of birth control include:

* Established use of oral, injected, or implanted hormonal methods of contraception that have comparable efficacy (failure rate < 1 %), for example hormone vaginal ring or transdermal hormone contraception
* Placement of an intrauterine device or intrauterine system
* Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of CAR001 for Phase I part | 4 weeks after last dosing of CAR001
  MTD was determined by testing increasing doses once a week for 4 weeks via IV on dose escalation cohorts 1 to 5 with 3 to 6 participants each. MTD reflects the highest dose of drug that did not cause a Dose-Limiting Toxicity (DLT) in > 33% of participants. DLTs were defined as any AE ≥ grade 3 (CTCAE v5.0) that is considered to be causally related (possibly, probably, or definitely related) to CAR001 within 4 weeks.
Objective Response Rate (ORR) of CAR001 for Phase IIa part | from visit 1 to 24-months of safety and efficacy follow-up period
  The rate of subjects with CR or PR based on RECIST1.1 in patients with NSCLC, TNBC or CRC; RANO in patients with GBM. Although there is no control group in this study, the ORR after CAR001 administration could be compared to baseline.

SECONDARY OUTCOMES:
Safety - AEs and SAEs incidences over the study period | from visit 1 to 24-months of safety and efficacy follow-up period
  The incidence of AEs and SAE from screening to the end of study or until documented disease progression.
Safety - Vital signs assessments at each post-treatment | from visit 1 to 24-months of safety and efficacy follow-up period
  Changes of vital signs at each post-treatment measurement or until documented disease progression from baseline.
Safety - Laboratory examinations at each post-treatment | from visit 1 to 24-months of safety and efficacy follow-up period
  Changes of laboratory data at each post-treatment measurement or until documented disease progression from baseline.
Safety - 12-lead electrocardiogram (ECG) assessments at each post-treatment | from visit 1 to 24-months of safety and efficacy follow-up period
  Changes of ventricular rate, PR interval, QRS interval, and QT interval by 12-lead ECG at each post-treatment measurement or until documented disease progression from baseline.
Safety - Physical Examination at each post-treatment | from visit 1 to 24-months of safety and efficacy follow-up period
  Abnormality in physical examination at each post-treatment measurement or until documented disease progression from baseline.
Efficacy - Progression Free Survival (PFS) rate | from visit 1 to 24-months of safety and efficacy follow-up period
  Time from 1st CAR001 administration to disease progression determined by MRI or CT, or death of the subject whichever comes first. Subjects who do not occur disease progression or mortality until the EOS will be considered as right-censored. Although there is no control group in this study, the PFS after CAR001 administration could be compared to historical data.
Efficacy - Overall Survival (OS) rate | from visit 1 to 24-months of safety and efficacy follow-up period
  Time from 1st CAR001 administration to death. Subjects who do not die until the end of study will be considered as right-censored. Although there is no control group in this study, the OS after CAR001 administration could be compared to historical data. After the EOS, the OS should be followed every 3 months by phone contact.
Efficacy - Change of QoL from baseline | from visit 1 to 24-months of safety and efficacy follow-up period
  QoL will be assessed by EORTC QLQ-C30 version 3.0 from baseline to subsequent evaluation visits or until documented disease progression.
Efficacy - Change of ECOG Performance Status Scale | from visit 1 to 24-months of safety and efficacy follow-up period
  ECOG Performance Status Scale will be assessed from baseline to subsequent evaluation visits or until documented disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Liang Huang, MD, Study Chair — Ever Supreme Bio Technology Co., Ltd.
Locations (1):
- China Medical University Hospital, Taichung, Non-US, Taiwan

REFERENCES:
- [Background] Huang SW, Pan CM, Lin YC, Chen MC, Chen Y, Jan CI, Wu CC, Lin FY, Wang ST, Lin CY, Lin PY, Huang WH, Chiang YT, Tsai WC, Chiu YH, Lin TH, Chiu SC, Cho DY. BiTE-Secreting CAR-gammadeltaT as a Dual Targeting Strategy for the Treatment of Solid Tumors. Adv Sci (Weinh). 2023 Jun;10(17):e2206856. doi: 10.1002/advs.202206856. Epub 2023 Apr 20. PMID 37078788